CLINICAL TRIAL: NCT06873867
Title: A Comparative Analysis in Treatment of Full-Thickness Wounds: NPWT Combined With Type-I Collagen Based Advanced Skin Substitute Versus NPWT Alone
Brief Title: Treatment of Full-Thickness Wounds: NPWT Combined With Type-I Collagen Based Advanced Skin Substitute Versus NPWT Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adichunchanagiri Institute of Medical Sciences, B G Nagara (Other)
Responsible Party: Principal Investigator, Dr Naveen Narayan MS, MCh (Plastic Surgery), Professor & HoD, Department of Plastic Reconstructive & Aesthetic Surgery, Adichunchanagiri Institute of Medical Sciences, B G Nagara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIMS/IEC/013/2025
Record Dates: First submitted 2025-03-03; First posted 2025-03-13 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Full Thickness Skin Defects; Ulcer
Keywords: Full Thickness Skin Defects; Ulcer; Negative Pressure Wound Therapy; High Purity Type 1 Collagen; Helicoll
MeSH Terms: conditions — Ulcer | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High Purity Type-I Collagen based Skin Substitute with Negative Pressure Wound Therapy (Active Comparator): In this study arm, wound is covered with High Purity Type-I Collagen (HPTC) based Skin Substitute applied followed by non adherent porous dressing followed by Negative Pressure Wound Therapy application set at 125mm of Hg pressure for 7 days. Procedure will be redone in case of need.
  Interventions: Device: High Purity Type-I Collagen based Skin Substitute; Device: Negative Pressure Wound Therapy
- Negative Pressure Wound Therapy (Active Comparator): In this study arm, wound is covered with non adherent porous dressing followed by Negative Pressure Wound Therapy application alone. Pressure is set at 125mm of Hg for 7 days. Procedure will be redone in case of need.
  Interventions: Device: Negative Pressure Wound Therapy

INTERVENTIONS:
Device: High Purity Type-I Collagen based Skin Substitute — In this wound care is covering with High Purity Type-I Collagen based Skin Substitute followed by a layer of non-adherent and porous dressing. After 5-7 days, wound examined and procedure is repeated as needed
  Arms: High Purity Type-I Collagen based Skin Substitute with Negative Pressure Wound Therapy
Device: Negative Pressure Wound Therapy — In this wound care is by application of Negative Pressure Wound Therapy using a standard polyurethane foam. The NPWT will be removed after 5-7 days, wound examined and procedure is repeated as needed

SUMMARY:
Widely used NPWT has been shown to promote wound healing by applying sub-atmospheric pressure, reducing oedema, and enhancing granulation tissue formation thus enhancing wound healing. However, its efficacy can vary based on wound characteristics and patient factors. High Purity Type-I Collagen (HPTC) based advanced skin substitute has emerged as a potential alternative for wound management, accelerating wound healing through extracellular matrix support. This study aims to compare the efficacy of NPWT combined with HPTC versus NPWT alone in the treatment of full-thickness wounds.

DETAILED DESCRIPTION:
Full-thickness wounds, extending through the dermis and affecting underlying tissues, present significant clinical challenges due to their complexity and prolonged healing times. Traditional treatments include surgical debridement, dressings, and advanced therapies like Negative Pressure Wound Therapy (NPWT). Widely used NPWT has been shown to promote wound healing by applying sub-atmospheric pressure, reducing oedema, and enhancing granulation tissue formation thus enhancing wound healing. However, its efficacy can vary based on wound characteristics and patient factors. High Purity Type-I Collagen (HPTC) based advanced skin substitute has emerged as a potential alternative for wound management, accelerating wound healing through extracellular matrix support. Studies suggest that HPTC promote cellular proliferation and angiogenesis, essential for tissue regeneration. Given the distinct mechanisms of action of NPWT and HPTC, a comparative evaluation is warranted to determine their relative efficacy in treating full-thickness wounds. This study aims to compare the efficacy of NPWT combined with HPTC versus NPWT alone in the treatment of full-thickness wounds.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age or older.
2. Presence of a full-thickness wound of at least 4 cm² and no more than 100 cm².
3. Wound duration of at least 4 weeks but not exceeding 6 months of standard of care prior to the initial screening visit.
4. Adequate vascular supply to the affected area
5. If the subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
6. The subject must agree to attend the twice-weekly/weekly study visits required by the protocol.
7. The subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

1. A subject known to have a life expectancy of <6 months
2. Wounds with active infection / osteomyelitis requiring systemic antibiotics.
3. Presence of malignancy in the wound bed.
4. Patients with uncontrolled diabetes (HbA1c > 9%).
5. Use of immunosuppressive therapy or systemic corticosteroids.
6. Use of other advanced wound care products within the past 30 days
7. Known allergy to fish products or components of HPTC.
8. Pregnant or breastfeeding women.
9. Presence of osteomyelitis or exposed bone, probes to bone or joint capsule on investigator's exam or radiographic evidence.
10. A subject receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent) or cytotoxic chemotherapy.
11. A subject with autoimmune or connective tissue disorders.
12. A subject who participated in a clinical trial involving treatment with an investigational product within the previous 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prema Dhanraj, MS, MCh, Study Chair — Rajarajeshwari Medical College and Hospital
Locations (1):
- Adichunchanagiri Institute of Medical Sciences, Mandya, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong DG, Lavery LA, Boulton AJ. Negative pressure wound therapy via vacuum-assisted closure following partial foot amputation: what is the role of wound chronicity? Int Wound J. 2007 Mar;4(1):79-86. doi: 10.1111/j.1742-481X.2006.00270.x. PMID 17425550
- [Background] Lee SK, An YS, Choy WS. Management of Hardware-Exposed Soft Tissue Defects Using Dermal Substitutes and Negative Pressure Wound Therapy. Ann Plast Surg. 2023 Mar 1;90(3):242-247. doi: 10.1097/SAP.0000000000003440. PMID 36796046
- [Background] Zhang L, Weng T, Wu P, Li Q, Han C, Wang X. The Combined Use of Negative-Pressure Wound Therapy and Dermal Substitutes for Tissue Repair and Regeneration. Biomed Res Int. 2020 Dec 4;2020:8824737. doi: 10.1155/2020/8824737. eCollection 2020. PMID 33344649
- [Background] Dhanraj P, Naveen N, Babu KR, Mahesh MS Hanumanthaiah KS. Healicoll: An Alternate to Flap Cover for Bare Bones and Tendons. Acta Medica International, 2016; 3(1): 146-150
- [Background] Narayan N, Gowda S, Shivannaiah C. A Randomized Controlled Clinical Trial Comparing the Use of High Purity Type-I Collagen-Based Skin Substitute vs. Dehydrated Human Amnion/Chorion Membrane in the Treatment of Diabetic Foot Ulcers. Cureus. 2024 Dec 5;16(12):e75182. doi: 10.7759/cureus.75182. eCollection 2024 Dec. PMID 39649230

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Purity Type-I Collagen Based Skin Substitute With Negative Pressure Wound Therapy | Negative Pressure Wound Therapy
Started | 52 | 52
Completed | 52 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Purity Type-I Collagen Based Skin Substitute With Negative Pressure Wound Therapy | Negative Pressure Wound Therapy | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Customized [Mean (Standard Deviation); unit: years] — Patients aged 18-80 years
  years | 54.1 (12.2) | 55.3 (11.7) | 54.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 34 | 33 | 67
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  India | 52 | 52 | 104
Wound area (cm²) [Mean (Standard Deviation); unit: square centimeters] | 32.8 (18.5) | 33.6 (17.9) | 33.18 (18.11)
Wound duration (weeks) [Mean (Standard Deviation); unit: weeks] | 4.1 (2.9) | 5.1 (3.1) | 4.6 (3.0)
Wound etiology, n (%) [Count of Participants; unit: Participants]
  Traumatic | 12 | 14 | 26
  Surgical | 10 | 10 | 20
  Diabetic | 8 | 10 | 18
  Burns | 8 | 8 | 16
  Vascular | 7 | 5 | 12
  Pressure | 7 | 5 | 12
Wound location, n (%) [Count of Participants; unit: Participants]
  Lower Limb | 28 | 23 | 51
  Chest | 10 | 9 | 19
  Upper limb | 8 | 12 | 20
  Abdomen | 4 | 5 | 9
  Back | 2 | 3 | 5
  Head and Neck | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Wound Area
Description: Percentage change in wound area from week 1 through week 7 measured manually with digital photography
Time Frame: 7 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | High Purity Type-I Collagen Based Skin Substitute With Negative Pressure Wound Therapy | Negative Pressure Wound Therapy
Number analyzed (Participants) | 52 | 52
percentage change
  Wound area reduction at 1 week | 23.73 (11.45) | 15.21 (9.32)
  Wound area reduction at 2 weeks | 34.47 (13.28) | 22.52 (10.85)
  Wound area reduction at 3 weeks | 45.17 (14.67) | 29.85 (11.98)
  Wound area reduction at 4 weeks | 56.45 (15.82) | 36.62 (12.74)
  Wound area reduction at 5 weeks | 67.14 (16.45) | 43.97 (13.28)
  Wound area reduction at 6 weeks | 78.33 (16.98) | 50.83 (13.72)
  Wound area reduction at 7 weeks | 89.35 (16.08) | 57.85 (12.73)

2. Secondary Outcome: Histopathological Analysis on Day 5 of Study
Description: Histopathological assessment will be done using biopsy on Day 0 of application to be compared with Day 5 after application of Type-I Collagen-based Skin Substitute or Human Amnion/Chorion Membrane. Histopathology assessed at day 0 and day 5, day 5 reported. Subsequently histopathology of biopsy will be done to look for:
  vascular infiltration (0-3 scale) - higher score means better, neo-epithelialization (0-3 scale) - higher score means better, fibroblast activity (0-3 scale) - higher score means better, inflammatory response (0-3 scale) - lower score means better and collagen deposition (0-3 scale) - higher score means better
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Purity Type-I Collagen Based Skin Substitute With Negative Pressure Wound Therapy | Negative Pressure Wound Therapy
Number analyzed (Participants) | 52 | 52
score on a scale
  vascular infiltration (0-3 scale) | 2.82 (0.65) | 2.10 (0.58)
  neo-epithelialization (0-3 scale) | 2.73 (0.61) | 1.72 (0.54)
  fibroblast activity (0-3 scale) | 2.79 (0.68) | 1.63 (0.52)
  inflammatory response (0-3 scale) | 1.32 (0.48) | 2.35 (0.63)
  collagen deposition (0-3 scale) | 2.78 (0.64) | 1.43 (0.49)

3. Secondary Outcome: Histopathological Analysis on Day 5 of Study - Capillary Density
Description: Histopathological assessment will be done using biopsy on Day 0 of application to be compared with Day 5 after application of Type-I Collagen-based Skin Substitute or Human Amnion/Chorion Membrane. Histopathology assessed at day 0 and day 5, day 5 reported. Subsequently histopathology of biopsy will be done to look for capillary density (vessels per mm²) - higher count means better,
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: vessels per mm²
Arm/Group | High Purity Type-I Collagen Based Skin Substitute With Negative Pressure Wound Therapy | Negative Pressure Wound Therapy
Number analyzed (Participants) | 52 | 52
vessels per mm² | 48.51 (8.32) | 42.97 (7.85)

4. Secondary Outcome: Time to Achieve Complete Wound Closure
Description: The time to achieve complete wound closure of the target ulcer by the end of 7 weeks
Time Frame: 7 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | High Purity Type-I Collagen Based Skin Substitute With Negative Pressure Wound Therapy | Negative Pressure Wound Therapy
Number analyzed (Participants) | 52 | 52
days | 36.81 (12.88) | 43.94 (16.70)

5. Secondary Outcome: Percentage of Participants to Obtain Complete Wound Closure
Description: The percentage of participants that obtain complete wound closure over the 7 weeks (6 weeks treatment period plus 1 week follow up)
Time Frame: 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High Purity Type-I Collagen Based Skin Substitute With Negative Pressure Wound Therapy | Negative Pressure Wound Therapy
Number analyzed (Participants) | 52 | 52
Participants | 45 | 22

6. Secondary Outcome: Percentage of Participants Achieving ≥50% Wound Healing
Description: Measurement of percentage of participants achieving ≥50% wound healing (epithelialization) assessed at follow up
Time Frame: 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High Purity Type-I Collagen Based Skin Substitute With Negative Pressure Wound Therapy | Negative Pressure Wound Therapy
Number analyzed (Participants) | 52 | 52
Participants | 49 | 27

7. Secondary Outcome: Mean Number of Application
Description: Mean number of rapplications of the NPWT+HPTC & NPWT alone used to obtain wound closure
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: number of applications
Arm/Group | High Purity Type-I Collagen Based Skin Substitute With Negative Pressure Wound Therapy | Negative Pressure Wound Therapy
Number analyzed (Participants) | 52 | 52
number of applications | 1.83 (0.82) | 4.3 (1.72)

8. Secondary Outcome: Number of Adverse Events
Description: Number of adverse events related to the intervention (e.g., infection, allergic reactions, NPWT seal issues)
Time Frame: 6 weeks
Measure: Number; unit: number of adverse events
Arm/Group | High Purity Type-I Collagen Based Skin Substitute With Negative Pressure Wound Therapy | Negative Pressure Wound Therapy
Number analyzed (Participants) | 52 | 52
number of adverse events
  Superficial wound infection | 2 | 3
  Skin irritation around wound | 1 | 1
  NPWT seal issues | 1 | 2
  Allergic reaction | 1 | 0
  Pain during dressing change | 0 | 2
  Severe infection requiring IV antibiotics | 0 | 0

9. Secondary Outcome: Pain Score on Visual Analog Scale
Description: Pain measured by a Visual Analog Scale with score range from 0 to 10, wherein 0="no pain" to 10="severe pain"
Time Frame: 7 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | High Purity Type-I Collagen Based Skin Substitute With Negative Pressure Wound Therapy | Negative Pressure Wound Therapy
Number analyzed (Participants) | 52 | 52
scores on a scale
  Baseline | 7.38 (1.85) | 7.16 (1.92)
  Week 1 | 6.36 (1.78) | 6.42 (1.82)
  Week 2 | 5.71 (1.72) | 5.97 (1.85)
  Week 3 | 4.73 (1.68) | 5.37 (1.79)
  Week 4 | 3.98 (1.62) | 4.94 (1.75)
  Week 5 | 2.86 (1.58) | 4.28 (1.72)
  Week 6 | 1.96 (1.52) | 3.83 (1.68)
  Week 7 | 1.51 (1.48) | 3.17 (1.65)

10. Secondary Outcome: Healed Wound Appearance Assessment Using Vancouver Scar Scale
Description: The resultant new skin is assessed and documented at each visit using the Vancouver Scar Scale, up to 7 weeks, week 7 visit reported, assessing vascularity, pigmentation, pliability and height/thickness with total score ranging from 0 to 13 (lesser the score better the scar)
Time Frame: 7 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | High Purity Type-I Collagen Based Skin Substitute With Negative Pressure Wound Therapy | Negative Pressure Wound Therapy
Number analyzed (Participants) | 52 | 52
scores on a scale | 3.9 (1.8) | 9.2 (2.5)

11. Secondary Outcome: Quality of Life Assessment
Description: The EuroQol 5-Dimension 5-Level (EQ-5D-5L) instrument is a standardized patient-reported outcome measure assessing overall health-related quality of life. It evaluates five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Scoring and Ranges:
  1. EQ-5D-5L Index Score - Derived from the five dimensions with five levels each (1 = no problems; 5 = extreme problems).
     The index score range varies by population value set; for most countries the possible scoring range is approximately -0.594 to 1.000. Higher scores indicate better health status (1.000 = full health).
  2. EQ Visual Analogue Scale (EQ-VAS) - A self-rated health scale from 0 to 100, where, 0 = the worst health you can imagine, 100 = the best health you can imagine. Higher values reflect better outcomes.
  Interpretation:
  Higher scores on both the EQ-5D-5L Index and EQ-VAS represent improved quality of life and a better treatment outcome.
Time Frame: 7 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | High Purity Type-I Collagen Based Skin Substitute With Negative Pressure Wound Therapy | Negative Pressure Wound Therapy
Number analyzed (Participants) | 52 | 52
scores on a scale
  EQ-5D Index Score | 0.91 (0.102) | 0.71 (0.116)
  EQ-VAS (0-100) | 88.2 (8.3) | 72.1 (9.0)

ADVERSE EVENTS:
Time Frame: 6-week treatment period + 1-week follow-up. Total 7 weeks
Description: All the study participants were considered at risk for adverse events.
Arm/Group | High Purity Type-I Collagen Based Skin Substitute With Negative Pressure Wound Therapy | Negative Pressure Wound Therapy
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 5/52 | 8/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Purity Type-I Collagen Based Skin Substitute With Negative Pressure Wound Therapy (N=52) | Negative Pressure Wound Therapy (N=52)
Superficial wound infection (Skin and subcutaneous tissue disorders) | 2 | 3
Skin irritation around wound (Skin and subcutaneous tissue disorders) | 1 | 1
NPWT seal issues (Product Issues) | 1 | 2
Allergic reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pain during dressing change (Skin and subcutaneous tissue disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
The single-center design may limit generalizability.

Complete blinding was not feasible due to the nature of interventions, potentially introducing bias, although outcome assessor blinding was maintained.

The 7-week study period, while adequate for assessing acute healing outcomes, may not capture long-term benefits or complications such as recurrence rates, functional outcomes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT06873867/Prot_SAP_003.pdf